CLINICAL TRIAL: NCT02112214
Title: Effect of Helicobacter Pylori Eradication on Gastric Cancer Prevention in Korea: a Randomized Controlled Clinical Trial
Brief Title: Helicobacter Pylori Eradication for Gastric Cancer Prevention in the General Population
Acronym: HELPER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: International Agency for Research on Cancer (Other); Chonnam National University Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Pusan National University Hospital (Other); Kyungpook National University Hospital (Other); Uijeongbu St. Mary's Hospital/The Catholic University (Unknown); Kangdong Sacred Heart Hospital (Other); Incheon St.Mary's Hospital/The Catholic University (Unknown); SMG-SNU Boramae Medical Center (Other); Chuncheon Sacred Heart Hospital (Other); Kosin University Gospel Hospital (Other)
Responsible Party: Principal Investigator, Il Ju Choi, Head of Gastric Cancer Cencer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NCCCTS13716; 1311240 (Other Grant/Funding Number: National Cancer Center, Korea)
Record Dates: First submitted 2014-04-03; First posted 2014-04-11 (Estimated); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Gastric Cancer; Helicobacter Pylori Infection
Keywords: Helicobacter pylori treatment; Gastric cancer; Screening
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Active Comparator): 10-day bismuth-based quadruple therapy for H. pylori positive subjects
  Interventions: Drug: 10-day bismuth-based quadruple therapy
- Placebo group (Placebo Comparator): Placebo for H. pylori positive subjects
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 10-day bismuth-based quadruple therapy — Bismuth 300 mg (4 times a day), lansoprazole 30 mg (twice a day), metronidazole 500 mg (3 times a day), and tetracycline 500 mg (4 times a day) for 10 days
  Other Names: Bismuth-based quadruple therapy
  Arms: Intervention group
Other: Placebo — Placebo for bismuth-based quadruple therapy
  Arms: Placebo group

SUMMARY:
The aim of this study is to define the role of H. pylori eradication in the prevention of gastric cancer and its precursors in the context of a population-based endoscopic screening program.

DETAILED DESCRIPTION:
Despite the decreasing incidence observed in the US and West European countries, gastric cancer is still an important global public health problem, especially in East Asian countries, where the burden of the disease is substantial. In the Republic of Korea, gastric cancer remains the leading cause of cancer in men and the fourth most common cancer in women. There is sufficient epidemiological and experimental evidence supporting a causal link between bacterial infection with H. pylori and gastric cancer development. However, evidence from clinical trials on the efficacy of H. pylori eradication with antimicrobial therapy to reduce the risk of gastric cancer is still limited. In addition, the beneficial or deleterious health impact of mass eradication at the population level has not been defined. In Korea, the prevalence of H. pylori infection in adults is still relatively high (~60%, >16 years old), and despite important reductions in mortality attributed to the screening program, incidence of gastric cancer remains elevated.

The investigators propose to conduct a randomized controlled clinical trial in Korea to evaluate the efficacy of H. pylori eradication to prevent gastric cancer incidence in different population subgroups including age and baseline gastric pathology. This study will be conducted in the context of the National Cancer Screening Program and the Korean Central Cancer Registry.

The proposed study will be a collaborative investigation between the National Cancer Center, Korea and the International Agency for Research on Cancer of the World Health Organization.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40-65 who are invited to participate in the National Cancer Screening Program and receive upper endoscopy
* Willingness to sign an informed consent form
* Good health, as determined by medical history and physical examination at enrollment

Exclusion Criteria:

* Personal history of gastric cancer
* Family history of gastric cancer in a first degree relative
* Diagnosis and active treatment for other organ cancer except carcinoma in situ within 5 years
* Current treatment for serious medical condition which could hinder participation (such as liver cirrhosis, renal failure, pulmonary dysfunction including COPD or asthma, or uncontrolled infection)
* Inadequate cardiovascular function including (a) New York Heart Association class III or IV heart disease, (b) unstable angina or myocardial infarction history, (c) history of significant ventricular arrhythmia requiring medication with antiarrhythmics, and (d) history of cerebrovascular accident
* Requirement for therapeutic anticoagulant therapy, aspirin
* Gastric resections due to benign disease
* H. pylori eradication therapy history
* Mental incompetence to understand and sign informed consent
* Alcoholism, drug abuse
* Serious chronic diseases according to the evaluation of the study physician
* Presence of a contraindication to the use of eradication treatment regimens
* Inability to provide an informed consent
* Pregnant or lactating women
* Treatment required due to peptic ulcer, gastric cancer or esophageal cancer identified during the endoscopic examination

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5224 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of gastric cancer between the intervention and placebo groups | Up to 10 years After H. pylori eradication
  Histologically confirmed gastric adenocarcinoma stage 1A or more advanced defined at endoscopy or through cancer registry

SECONDARY OUTCOMES:
Incidence of gastric dysplasia | Up to 10 years After H. pylori eradication
  Diagnosis of histologically confirmed gastric dysplasia
Occurrence of adverse events caused by antibiotic treatment | During 10 days of H. pylori eradication, and Up To 1 month after the treatment completion
  Solicited/unsolicited adverse events
Incidence and mortality from other medical conditions such as obesity, diabetes, circulatory diseases, oesophageal diseases as well as other cancers and cognitive impairment | Up to 10 years After H. pylori eradication
  Assessed through record linkage or direct assessment during screening visits
Mortality from gastric cancer | Up to 10 years after eradication
  Cancer registry or other reports
All-cause mortality | Up to 10 years After H. pylori eradication
  Korean National Health Insurance records or other reports
Modification of atrophy score | Up to 10 years After H. pylori eradication
  Change in histologic atrophy grade from enrollment to subsequent endoscopic assessment

CONTACTS AND LOCATIONS:
Overall Officials: Il Ju Choi, M.D., Ph.D., Study Director — National Cancer Center, Korea; Rolando Herrero, M.D.,Ph.D, Principal Investigator — International Agency for Research on Cancer
Locations (11):
- South Korea (11):
  - Kosin University Gospel Hospital, Busan
  - Pusan National University Hospital, Busan
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon
  - Kyungpook National University Hospital, Daegu
  - National Cancer Center, Goyang
  - Chonnam National University Hospital, Gwangju
  - Incheon St.Mary's Hospital/The Catholic University, Incheon
  - Kandong Sacred Heart Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Uijeongbu St. Mary's Hospital/The Catholic University, Uijeongbu-si